CLINICAL TRIAL: NCT04022278
Title: Evaluation of the Population Likely to Benefit From Sleep Exploration: Cross-sectional Study on a Given Day Within the Paris Saint-Joseph Hospital Group
Brief Title: Cross-sectional Study on a Given Day Within the Paris Saint-Joseph Hospital Group
Acronym: EXPLOSOM
Status: Withdrawn | Type: Observational
Why Stopped: The PI decided it.
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: EXPLOSOM
Record Dates: First submitted 2019-07-15; First posted 2019-07-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sleep apnea syndrome has an estimated incidence of 2 to 4% in the adult population and more so in men and with aging. It is an independent risk factor for mortality. Cardiovascular pathologies, diabetes, and stroke are known comorbidities with a high rate of association. There is no recommendation to screen these patients although the interest is assumed and sleep apnea syndrome is largely underdiagnosed. Interrogation and clinical examination guide but they are neither sensitive nor specific. The use of scores improves screening. In the general population, the Berlin score has a high false negative rate. The STOP-BANG score is sensitive but with a poor positive predictive value. Combined, these scores can be used to detect Sleep Apnea Syndrome. The interest of a management was especially shown for the very symptomatic syndromes because it is a pledge of observance of the treatment, itself necessary for the effectiveness in the prevention of the cardiovascular complications.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is> 18 years
* Any patient hospitalized on the day of the survey in any of the services of the cardio-neurovascular division of the Paris Saint-Joseph Hospital Group, whatever the history of comorbidities, the reason for hospitalization
* Francophone patient

Exclusion Criteria:

* Patient under tutorship or curatorship
* Patient deprived of liberty
* Patient at the end of life
* Patient opposing his participation in the research protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient hospitalized on the day of the survey in any of the services of the cardio-neurovascular division of the Paris Saint-Joseph Hospital Group, whatever the history of comorbidities, the reason for hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

PRIMARY OUTCOMES:
Patients with severe co-morbidities whose clinical presentation suggests sleep apnea syndrome sufficiently severe and symptomatic to benefit from sleep exploration | Day 1
  This outcome measure the roportion of patients with all of the criteria defining the patient as "comorbid and symptomatic suspect".

CONTACTS AND LOCATIONS:
Overall Officials: Claire P GAZANIOL, MD, Principal Investigator — Fondation Hôpital Saint-Joseph